CLINICAL TRIAL: NCT01199146
Title: A Phase II Study of Abiraterone Acetate in Patients With Castration Resistant Prostate Cancer (CRPC) and Prior Therapy With Ketoconazole
Brief Title: Abiraterone Post Ketoconazole for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Johnson & Johnson (Industry); Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC# 085514
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-12

CONDITIONS: Prostate Cancer
Keywords: Abiraterone acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abiraterone acetate (Experimental)
  Interventions: Drug: Abiraterone acetate

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate 1000 mg by mouth per day
  Other Names: CB7630

SUMMARY:
This is a phase II, open label, single center study to evaluate the efficacy of abiraterone acetate (CB7630) administered to patients with castrate resistant prostate cancer who have experienced disease progression on ketoconazole.

It is hypothesized that abiraterone will be active in patients who have experienced disease progression on ketoconazole

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Prior therapy with ketoconazole for castration resistant prostate cancer. Patients should demonstrate evidence of progression (see below definitions) on ketoconazole or evidence of grades 3/4 toxicities on ketoconazole.

  1. Ketoconazole must have been administered for >28 days
  2. At least 27 days must elapse since last ketoconazole dose and first dose of abiraterone acetate
* No prior therapy with chemotherapy for metastatic prostate cancer
* Metastatic disease based on a positive bone scan or objective imaging on CT scan
* Ongoing gonadal androgen deprivation therapy with LHRH analogues or orchiectomy. Patients, who have not had an orchiectomy, must be maintained on effective LHRH analogue therapy for the duration of the trial
* Testosterone < 50 ng/dL
* Progressive disease after androgen deprivation: PSA evidence for progressive prostate cancer consists of a PSA level of at least 2 ng/ml which has risen on at least 2 successive occasions, at least 2 weeks apart
* Patients who are receiving an antiandrogen as part of primary androgen ablation must demonstrate disease progression following discontinuation of antiandrogen
* ECOG Performance Status 0-1
* Age >18 years and able to comply with protocol requirements
* Serum Creatinine ≤1.5 x ULN
* Serum potassium >3.5mmol/L
* Bilirubin ≤1.5x ULN
* AST and ALT ≤2.5 x ULN
* Life expectancy of >12 weeks

Exclusion Criteria:

* Therapy with other hormonal therapy, including any dose of megestrol acetate (Megace), finasteride (Proscar), dutasteride (Avodart) any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES), or any systemic corticosteroid within 4 weeks prior to first dose of study drug
* Therapy with supplements or complementary medicines/botanicals within 4 weeks of first dose of study drug, except for any combination of the following; conventional multivitamin supplements, Selenium, Lycopene and Soy supplements
* Prior radiation therapy completed < 4 weeks prior to enrollment
* Prior chemotherapy for castration resistant prostate cancer. Patients who have received chemotherapy for early stage prostate cancer (e.g. as part of a neoadjuvant or adjuvant trial) or for other malignancies are eligible provided that >1 year has passed since the administration of the last chemotherapy dose.
* Hemoglobin ≤9.0 g/dL
* Any "currently active" second malignancy, other than non-melanoma skin cancer Patients are not considered to have a "currently active" malignancy, if they have completed therapy and are considered by their physician to be at least less than 30% risk of relapse over next 3 months
* Blood pressure that is not controlled despite >2 oral agents (SBP >160 and DBP >90 on three or more readings within the screening period)
* Serum K+ <3.5 mmoL/L on more than one reading within the screening period
* NYHA Class II, NYHA Class III or IV Congestive Heart Failure
* Myocardial infarction within the 6 months prior to the first dose of study drug
* Serious intercurrent infections or nonmalignant medical illnesses that are uncontrolled
* Concurrent therapy with drugs that are metabolized as substrates of CYP1A2, CYP2D6, or CYP2C19 and are considered by the investigators to pose a risk for drug to drug interactions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-09-10 (Actual); Primary Completion 2013-01-04 (Actual); Study Completion 2016-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Ryan, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Chicago, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abiraterone Acetate
Started | 42
Completed | 39
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 71 [59 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Preliminary Evidence of Efficacy of Abiraterone Acetate
Description: number of patients with ≥ 30% PSA decline after 12 weeks of abiraterone treatment
Time Frame: 12 weeks from beginning of abiraterone treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 39
Participants | 20

2. Secondary Outcome: Time To Progression (TTP)
Time Frame: beginning of treatment until disease progression according to Prostate Cancer Working Group 2 (PCWG2) criteria
Measure: Median (Full Range); unit: weeks
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 39
weeks | 16 [4 to 71]

3. Secondary Outcome: Proportion of Patients With PSA Decline of > 50%
Time Frame: 12 weeks from beginning of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 39
Participants | 19

ADVERSE EVENTS:
Arm/Group | Abiraterone Acetate
All-Cause Mortality (participants affected / at risk) | 2/42
Serious Adverse Events (participants affected / at risk) | 5/42
Other Adverse Events (participants affected / at risk) | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=42)
Hemoglobin (Blood and lymphatic system disorders) | 2
Constitutional Symptoms - Other (Specify, __) (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1
Weight loss (General disorders) | 1
Death not associated with CTCAE term - Sudden death (General disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Infection - Other (Specify, __) (Infections and infestations) | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Pain - Back (General disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=42)
Hemoglobin (Blood and lymphatic system disorders) | 13
Platelets (Blood and lymphatic system disorders) | 2
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1
Vasovagal episode (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 11
Hypotension (Cardiac disorders) | 1
Constitutional Symptoms - Other (Specify, __) (General disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 31
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2
Insomnia (General disorders) | 1
Sweating (diaphoresis) (General disorders) | 1
Weight gain (General disorders) | 2
Weight loss (General disorders) | 3
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 1
Death not associated with CTCAE term - Sudden death (General disorders) | 1
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 3
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 2
Flushing (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Hot flashes/flushes (Endocrine disorders) | 4
Anorexia (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 7
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Salivary gland changes/saliva (Gastrointestinal disorders) | 1
Infection - Other (Specify, __) (Infections and infestations) | 3
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1
Edema: head and neck (Blood and lymphatic system disorders) | 1
Edema: limb (Blood and lymphatic system disorders) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 5
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3
Alkaline phosphatase (Metabolism and nutrition disorders) | 8
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 6
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 7
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 18
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 2
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Mood alteration - Anxiety (Nervous system disorders) | 1
Mood alteration - Depression (Nervous system disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 1
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1
Uveitis (Eye disorders) | 3
Pain - Back (General disorders) | 9
Pain - Bone (General disorders) | 1
Pain - Buttock (General disorders) | 1
Pain - External ear (General disorders) | 1
Pain - Extremity-limb (General disorders) | 7
Pain - Eye (General disorders) | 1
Pain - Head/headache (General disorders) | 1
Pain - Joint (General disorders) | 4
Pain - Muscle (General disorders) | 4
Pain - Other (Specify, __) (General disorders) | 7
Pain - Pain NOS (General disorders) | 6
Pain - Pelvis (General disorders) | 8
Pain - Tumor pain (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1
Incontinence, urinary (Renal and urinary disorders) | 1
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No